CLINICAL TRIAL: NCT05445245
Title: The Longitudinal Study of Low Anterior Resection Syndrome, Psychological Distress, and Fecal Incontinence-related Quality of Life in Patients with Newly Diagnosed Rectal Cancer.
Brief Title: The Longitudinal Study of Low Anterior Resection Syndrome in Patients with Newly Diagnosed Rectal Cancer.
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202101979B0
Record Dates: First submitted 2022-06-30; First posted 2022-07-06 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-02

CONDITIONS: Rectal Cancer
Keywords: low anterior resection syndrome; psychological distress; quality of life; rectal cancer
MeSH Terms: conditions — Rectal Neoplasms; Low Anterior Resection Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aims are to identify the trajectory of LAR Syndrome and explore the adaptation process and coping strategies of LAR Syndrome in patients newly diagnosed with rectal cancer. The participants will recruit from a CRC surgical outpatient department of a medical center in northern Taiwan.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with stage I to III rectal cancer.
2. Patients already know their condition.

4. Aged 20 years and older. 5. Consciously communicate in Mandarin or Taiwanese. 6. Agreed with the interview and had signed the permit.

Exclusion Criteria:

1. Patients with Stage IV rectal cancer.
2. Recurred rectal cancer.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rectal cancer patients during therapy.
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-24 (Actual)

PRIMARY OUTCOMES:
Self-report Questionnaire | Change from baseline symptom at 12 months
  show the specific trajectory of LAR Syndrome, psychological distress, and fecal incontinence-related QoL based on different tumor locations in patients with rectal cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Chung Gung University, Taoyuan, Kwei-Shan Dist., Taiwan